CLINICAL TRIAL: NCT07324772
Title: PREACTIVE: Preconditioning With REsistance and AerobiC Training to ImproVe Exercise Intolerance and Quality of Life in Comorbid Atrial Fibrillation and HFpEF
Brief Title: PREACTIVE: Preconditioning Exercise Intervention to Improve Symptoms and Quality of Life in Comorbid Atrial Fibrillation and HFpEF
Acronym: PREACTIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Deepika Laddu, PI, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU#: 00223545
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation (Paroxysmal); Persistent Atrial Fibrillation; Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: exercise; exercise capacity; symptom severity; quality of life
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This single arm pilot study will recruit 30 patients aged ≥60 years with persistent AF and HFpEF for a 4-month PREACTIVE intervention. Participants will complete 16 weeks of exercise (3 sessions per week) with a study exercise interventionist (trainer). PREACTIVE comprises of two phases, each lasting 2 months (8 weeks, 3 sessions/week; 24 sessions total). Phase I employs progressive resistance training (PRT)-only to promote gains in muscle mass and strength, and neuromuscular function. Phase II includes 8 weeks (3 sessions/week; 24 sessions total) that will continue with an abbreviated version of PRT while focusing on aerobic endurance training. Aerobic training will gradually progress by workload and the heart rate reserve (HRR) method will be used to guide exercise intensity. The HRR is determined from the 6-minute walk test (6MWT) performed at the baseline visit and rate of perceived exertion (RPE) will be used to guide intensity and progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PREACTIVE (Experimental): During Phase I participants will engage first in progressive resistance training only (3 sessions/week; 24 sessions total) to optimize gains in muscle mass and strength, neuromuscular function, and hemodynamic gains. Phase II includes 8 weeks that focus on aerobic endurance training and also an abbreviated version of PRT (3 sessions/week; 24 sessions total).
  Interventions: Behavioral: progressive resistance training; Behavioral: combined aerobic + resistance training

INTERVENTIONS:
Behavioral: progressive resistance training — 2 months of progressive resistance training, performed for 3 sessions/week; 24 sessions total, under supervision with a trainer (1:1 interaction) Sessions include six upper- and lower-extremity exercises performed in alternate pattern as described (e.g., chest press, seated leg press, seated latissimus pull-down, knee/leg extension, shoulder press, leg curls) using pressurized or weighted machines. Participants will start the intensity of 40-50% of their baseline 1 repetition maximum (1-RM), with the goal of progressing to 70-80% of their 1-RM by 8 weeks, if able. Progression in intensity and reps will follow the principles of overload, such that resistance will be incremented only when a subject completes 12 reps for at least 2 of the 3 total sets at a given resistance, complemented by a reduction in the number of reps per set.
Behavioral: combined aerobic + resistance training — Phase II comprises of 8 weeks of aerobic training (primary focus) while continuing a shortened PRT protocol comprising of 3-4 exercises targeting upper and lower body. Sessions will be 3 sessions/week; 24 sessions total). Initial training intensity will be 40-50% of the HRR from the 6MWT with the goal of progressing to 60%-70% of HRR and for 20-35min over 8 weeks. Goals will be adjusted to 40%-50% HRR and 15-30min of exercise for those unable to meet targets.

SUMMARY:
Atrial fibrillation (AF) and heart failure with preserved ejection fraction (HFpEF) are very common conditions that often occur together and result in worsening symptoms and reduced quality of life (QoL). Limitations being able to participate in activities of daily living is a primary complaint for AF-HFpEF patients, yet effective strategies to address this issue remain limited. While exercise interventions targeting aerobic training (AT) are recommended for patients with AF and HFpEF, unique challenges exist in this patient population who tend to be older. Specifically, many older patients with AF and HFpEF have muscle weakness, sarcopenia and frailty, that can make aerobic-focused exercise difficult and less tolerable. This study proposes that starting with progressive resistance training (PRT) before aerobic exercise may overcome these issues by improving muscle strength, making AT more manageable, and leading to better health outcomes. The goal of this study is to assess whether a sequential exercise program, named 'PREACTIVE' improves how people feel, decrease the amount of symptoms, and their ability to participate in exercise and activities.

This study will specifically test a sequenced exercise approach of resistance training followed by aerobic exercise to improve symptoms, and quality of life in AF-HFpEF.

DETAILED DESCRIPTION:
The main objective of this research to evaluate the feasibility and preliminary efficacy of a pilot exercise training program ('PREACTIVE') sequenced specifically for optimal function in AF-HFpEF on aerobic capacity (primary outcome), and its relation to secondary measures-muscle strength, physical function, AF symptom burden and QoL.

ELIGIBILITY:
Inclusion Criteria:

All participants will be age 60 and older, have a primary diagnosis of AF and HFpEF, based on electronic health record review. Patients with persistent AF or Paroxysmal AF are eligible. HFpEF will be defined in accordance to the 2022 AHA/ACC/HFSA Guideline using a clinical composite score, the H2FPEF score, in conjunction with diagnostic criteria below:

* Ejection fraction ≥ 50%
* E/e' ≥15 by Doppler Echocardiography
* High H2FpEF score (≥5)
* Must be in stable medical condition and able to begin an exercise program

Exclusion Criteria:

* Valvular heart disease as the primary etiology of heart failure (i.e., severe aortic stenosis or mitral regurgitation),
* New York Heart Association Stage IV
* Recent stroke (<1 year)
* Evidence or History of Cardiac amyloidosis
* Patients with persistent AF and poor rate control (HR > 110 at rest)
* Significant change in cardiac medication or Heart Failure symptoms < 2 weeks
* Unstable or severe angina not controlled during daily activity by pharmacological therapy or at <4 METS activity
* Uncontrolled hypertension (defined as systolic blood pressure >200 mm Hg and/or diastolic blood pressure>110 mm Hg) with medications
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Hospitalization or urgent care visit < 4 weeks
* Oxygen dependent Chronic Obstructive Pulmonary Disease (COPD)
* Significant anemia (<10 g/dL Hgb)
* End stage renal replacement therapy associated with the need for dialysis
* Active treatment for cancer defined as current radiation, chemotherapy, immunotherapy, or cancer recurrence within past 5 years
* Hospice care and indication of life expectancy less than 2 years
* Complete dependence confinement to a Wheelchair confinement or requiring a visual impairment or Orthopedic or severe musculoskeletal conditions that would prohibit resistance training or aerobic exercise.
* Physician diagnosed Alzheimer's disease or Dementia or bipolar or psychotic disorder; Montreal Cognitive Assessment (MoCA) is ≤ 18 (based on participant screening)
* High levels of physical functioning based the composite short physical performance battery score of ≥10 (out of 12)
* Planned major surgery, coronary or leg revascularization during the next six months
* Participation in a supervised exercise program or already engaging in regular exercise
* Plans to transfer care outside of NU within the study period
* Unable to consent or commit to requires study procedures
* Non-English speaking

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test (4 month change) | change from baseline visit to 4 months (post intervention visit)
  Submaximal aerobic capacity by the 6-minute walk test [6MWT]

SECONDARY OUTCOMES:
muscle strength | change from baseline visit to 4 months (post-intervention visit)
  change in muscle strength assessed by 1-repetition maximum (or equivalent) for chest press and leg press
short physical performance battery | change from baseline to 4 months (post intervention visit)
  Physical function short physical performance battery
Atrial Fibrillation symptom severity by the Atrial Fibrillation Severity Scale (AFSS) | change from baseline to 4 months (post-intervention visit)
  Atrial Fibrillation symptom severity by the Atrial Fibrillation Severity Scale (AFSS)
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire | change from baseline to 4 months (post intervention visit)
  Afib specific quality of life
Kansas City Cardiomyopathy Questionnaire | change from baseline to 4 months (post intervention visit)
  overall (HF specific) health-related quality of life by the Kansas City Cardiomyopathy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Laddu, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No